CLINICAL TRIAL: NCT01330342
Title: Evolution of Cellular and Viral Resistance in HIV-infected Patients With Lymphoma
Acronym: SSAT042
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SSAT 042
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: HIV; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV patients without lymphoma: HIV-infected subjects on cART without a diagnosis of lymphoma
- HIV patients with lymphoma: HIV seropositive individuals with lymphoma

SUMMARY:
The study's chief objective is to observe the evolution of cellular (in terms of expression of transmembrane transporters and their transcriptional regulators) and viral resistance (in terms of development of mutations in the HIV genome that may confer resistance to future treatment for HIV) in HIV-infected patients with lymphoma.

DETAILED DESCRIPTION:
The study team will take two or three tubes of blood on three occasions during the course of chemotherapy. The total amount of blood required for this research project is 64mL (approximately 4 tablespoons).

This will allow better understanding of the changes that take place in the blood and the HIV virus itself. It is hoped that this will provide new insights that may aid the understanding and treatment of HIV patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
* Documented HIV-1 infection.
* Diagnosis of lymphoma (with the exclusion of the five subjects that will be controls).
* On cART or about to start cART as part of clinical routine care before the initiation of chemotherapy.

Exclusion Criteria:

- Receiving anti-tuberculosis treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV seropositive individuals with and without lymphoma.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Development of multi-drug resistance (in terms of expression of transmembrane transporters and their transcriptional regulators) in HIV-infected patients with lymphoma. | 3 years

SECONDARY OUTCOMES:
Development of mutations in the HIV genome that may confer resistance to future treatment for HIV. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom